CLINICAL TRIAL: NCT00000797
Title: Women's Interagency HIV Study (WIHS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: WIHS
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bodily fluid, and hair collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Women's Interagency HIV Study (WIHS), a multicenter, prospective study, was established in August 1993 to carry out comprehensive investigations of the impact of HIV infection and its clinical, laboratory, and psychosocial effects in women. The purpose of this study is to collect and evaluate these data from HIV infected and at-risk women to better understand and provide support for women whom are currently HIV infected or who are at risk for HIV infection.

DETAILED DESCRIPTION:
HIV in women is increasing worldwide, with women comprising approximately 14% of the total adult and adolescent AIDS cases, the highest proportion yet reported. The impact of AIDS is particularly severe in minority populations; among women, African Americans, and Hispanics combined now represent the majority of AIDS cases (76%) in the United States. AIDS is now the third leading cause of death for women aged 25 to 44 (after cancer and cardiovascular disease) and is the leading cause of death of African American women in this age group.

Studies of HIV and AIDS in women can play a unique role in testing new biological or socio-behavioral hypotheses at the population level and in linking basic science findings and laboratory methods to well-defined populations and communities. Research areas that are likely to draw more attention in the near future will include the study of pathogenicity and transmissibility of different HIV subtypes or recombinant forms and their interaction with variably susceptible individuals; the change in the scope of HIV natural history studies in the era of combination antiretroviral therapy; and the contribution of such studies to the design of a wide spectrum of prevention modalities (e.g., prevention of HIV and prevention of opportunistic infections). In addition, studies of natural history of HIV-related malignancies and active surveillance of malignancies in HIV infected and high-risk uninfected women may lead to new screening and prevention modalities in high-risk populations of women.

Participants will have study visits every 6 months. Questionnaires regarding sexual behavior, health care utilization, medical and obstetric/gynecological history, psychosocial factors, and sociodemographics will be completed by participants. Physical, gynecological, and lipodystrophy examinations will also be conducted at each visit, and current medication regimen will be noted. Blood and other bodily fluid samples will be collected and registered in both local and national repositories of the WIHS in conjunction with NIAID.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Willing to be retested for HIV infection for this study unless hardcopy documentation of a positive result (HIV ELISA test and a confirmatory Western blot) is available
* Either have never taken HIV antiretroviral medications or have a documented start date of highly active antiretroviral therapy (HAART) after January 1, 2008
* If have taken HAART, have documentation of pre-HAART CD4 counts and HIV RNA quantification
* Willing and able to have blood drawn
* Give consent to have their specimens stored in the WIHS national repository
* Able to complete study visit interviews in English or Spanish every 6 months
* Able to travel to and from site clinic and participate in study visits as an outpatient

Exclusion Criteria:

* Perinatally acquired HIV
* Enrolled in the WIHS through another site
* HAART started before January 1, 2008, except during pregnancy
* Participant plans to move out of the area within 12 months

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV-infected women and HIV-uninfected women who are at risk of HIV infection
Sampling Method: Probability Sample
Enrollment: 4982 (Estimated)
Dates: Start 1994-10; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California - San Francisco, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Chicago Consortium, Chicago, Illinois
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Massad LS, Riester KA, Anastos KM, Fruchter RG, Palefsky JM, Burk RD, Burns D, Greenblatt RM, Muderspach LI, Miotti P. Prevalence and predictors of squamous cell abnormalities in Papanicolaou smears from women infected with HIV-1. Women's Interagency HIV Study Group. J Acquir Immune Defic Syndr. 1999 May 1;21(1):33-41. doi: 10.1097/00126334-199905010-00005. PMID 10235512
- [Result] Anastos K, Kalish LA, Hessol N, Weiser B, Melnick S, Burns D, Delapenha R, DeHovitz J, Cohen M, Meyer W, Bremer J, Kovacs A. The relative value of CD4 cell count and quantitative HIV-1 RNA in predicting survival in HIV-1-infected women: results of the women's interagency HIV study. AIDS. 1999 Sep 10;13(13):1717-26. doi: 10.1097/00002030-199909100-00016. PMID 10509574
- [Result] Feldman JG, Burns DN, Gange SJ, Bacchetti P, Cohen M, Anastos K, Nowicki M, Delapena R, Miotti P. Serum albumin as a predictor of survival in HIV-infected women in the Women's Interagency HIV study. AIDS. 2000 May 5;14(7):863-70. doi: 10.1097/00002030-200005050-00013. PMID 10839595
- [Result] DeHovitz JA, Kovacs A, Feldman JG, Anastos K, Young M, Cohen M, Gange SJ, Melnick S, Greenblatt RM. The relationship between virus load response to highly active antiretroviral therapy and change in CD4 cell counts: A report from the Women's interagency HIV study. J Infect Dis. 2000 Nov;182(5):1527-30. doi: 10.1086/315875. Epub 2000 Sep 27. PMID 11010840
- [Result] Levine AM, Berhane K, Masri-Lavine L, Sanchez M, Young M, Augenbraun M, Cohen M, Anastos K, Newman M, Gange SJ, Watts H. Prevalence and correlates of anemia in a large cohort of HIV-infected women: Women's Interagency HIV Study. J Acquir Immune Defic Syndr. 2001 Jan 1;26(1):28-35. doi: 10.1097/00126334-200101010-00004. PMID 11176266
- [Result] Minkoff H, Ahdieh L, Watts H, Greenblatt RM, Schmidt J, Schneider M, Stek A. The relationship of pregnancy to the use of highly active antiretroviral therapy. Am J Obstet Gynecol. 2001 May;184(6):1221-7. doi: 10.1067/mob.2001.113871. PMID 11349192
- [Result] French AL, Kirstein LM, Massad LS, Semba RD, Minkoff H, Landesman S, Palefsky J, Young M, Anastos K, Cohen MH. Association of vitamin A deficiency with cervical squamous intraepithelial lesions in human immunodeficiency virus-infected women. J Infect Dis. 2000 Oct;182(4):1084-9. doi: 10.1086/315816. Epub 2000 Sep 1. PMID 10979903
- [Result] Greenspan D, Komaroff E, Redford M, Phelan JA, Navazesh M, Alves ME, Kamrath H, Mulligan R, Barr CE, Greenspan JS. Oral mucosal lesions and HIV viral load in the Women's Interagency HIV Study (WIHS). J Acquir Immune Defic Syndr. 2000 Sep 1;25(1):44-50. doi: 10.1097/00042560-200009010-00006. PMID 11064503
- [Result] Mirmirani P, Hessol NA, Maurer TA, Berger TG, Nguyen P, Khalsa A, Gurtman A, Micci S, Young M, Holman S, Gange SJ, Greenblatt RM. Prevalence and predictors of skin disease in the Women's Interagency HIV Study (WIHS). J Am Acad Dermatol. 2001 May;44(5):785-8. doi: 10.1067/mjd.2001.112350. PMID 11312425
- [Result] Stancliff S, Abel S, Agins B. Oral mucosal lesions and HIV viral load in the Women's Interagency HIV Study (WIHS). J Acquir Immune Defic Syndr. 2001 May 1;27(1):96-7. doi: 10.1097/00126334-200105010-00019. No abstract available. PMID 11404529
- [Result] Justman JE, Benning L, Danoff A, Minkoff H, Levine A, Greenblatt RM, Weber K, Piessens E, Robison E, Anastos K. Protease inhibitor use and the incidence of diabetes mellitus in a large cohort of HIV-infected women. J Acquir Immune Defic Syndr. 2003 Mar 1;32(3):298-302. doi: 10.1097/00126334-200303010-00009. PMID 12626890
- [Result] Kirstein LM, Greenblatt RM, Anastos K, Levine A, French AL, Minkoff H, Silver S, Gange SJ; Women's Interagency HIV Study Collaborative Research Group. Prevalence and correlates of highly active antiretroviral therapy switching in the Women's Interagency HIV Study. J Acquir Immune Defic Syndr. 2002 Apr 15;29(5):495-503. doi: 10.1097/00126334-200204150-00010. PMID 11981366
- [Result] Preston-Martin S, Kirstein LM, Pogoda JM, Rimer B, Melnick S, Masri-Lavine L, Silver S, Hessol N, French AL, Feldman J, Sacks HS, Deely M, Levine AM. Use of mammographic screening by HIV-infected women in the Women's Interagency HIV Study (WIHS). Prev Med. 2002 Mar;34(3):386-92. doi: 10.1006/pmed.2001.1003. PMID 11902857
- [Result] Mulligan R, Phelan JA, Brunelle J, Redford M, Pogoda JM, Nelson E, Seirawan H, Greenspan JS, Navazesh M, Greenspan D, Alves ME. Baseline characteristics of participants in the oral health component of the Women's Interagency HIV Study. Community Dent Oral Epidemiol. 2004 Apr;32(2):86-98. doi: 10.1111/j.0301-5661.2004.00128.x. PMID 15061857
- [Result] Strickler HD, Palefsky JM, Shah KV, Anastos K, Klein RS, Minkoff H, Duerr A, Massad LS, Celentano DD, Hall C, Fazzari M, Cu-Uvin S, Bacon M, Schuman P, Levine AM, Durante AJ, Gange S, Melnick S, Burk RD. Human papillomavirus type 16 and immune status in human immunodeficiency virus-seropositive women. J Natl Cancer Inst. 2003 Jul 16;95(14):1062-71. doi: 10.1093/jnci/95.14.1062. PMID 12865452
- [Result] Silverberg MJ, Ahdieh L, Munoz A, Anastos K, Burk RD, Cu-Uvin S, Duerr A, Greenblatt RM, Klein RS, Massad S, Minkoff H, Muderspach L, Palefsky J, Piessens E, Schuman P, Watts H, Shah KV. The impact of HIV infection and immunodeficiency on human papillomavirus type 6 or 11 infection and on genital warts. Sex Transm Dis. 2002 Aug;29(8):427-35. doi: 10.1097/00007435-200208000-00001. PMID 12172526
- [Result] Richardson JL, Martin EM, Jimenez N, Danley K, Cohen M, Carson VL, Sinclair B, Racenstein JM, Reed RA, Levine AM. Neuropsychological functioning in a cohort of HIV infected women: importance of antiretroviral therapy. J Int Neuropsychol Soc. 2002 Sep;8(6):781-93. doi: 10.1017/s1355617702860064. PMID 12240742
- [Result] Szczech LA, Gange SJ, van der Horst C, Bartlett JA, Young M, Cohen MH, Anastos K, Klassen PS, Svetkey LP. Predictors of proteinuria and renal failure among women with HIV infection. Kidney Int. 2002 Jan;61(1):195-202. doi: 10.1046/j.1523-1755.2002.00094.x. PMID 11786101
- [Result] Minkoff H, Ahdieh L, Massad LS, Anastos K, Watts DH, Melnick S, Muderspach L, Burk R, Palefsky J. The effect of highly active antiretroviral therapy on cervical cytologic changes associated with oncogenic HPV among HIV-infected women. AIDS. 2001 Nov 9;15(16):2157-64. doi: 10.1097/00002030-200111090-00011. PMID 11684935
- [Result] Augenbraun M, Tarwater P, Greenblatt R, Cohen M, French A, Gore ME, Watts H, Preston-Martin S, Anastos K; Women's Interagency HIV Study (WIHS). Opportunistic infection prophylaxis in the women's interagency HIV study (WIHS). J Acquir Immune Defic Syndr. 2001 Oct 1;28(2):195-6. doi: 10.1097/00126334-200110010-00014. No abstract available. PMID 11588516
- [Result] Hessol NA, Anastos K, Levine AM, Ameli N, Cohen M, Young M, Augenbraun M, Miotti P, Gange SJ. Factors associated with incident self-reported AIDS among women enrolled in the women's interagency HIV study (WIHS). WIHS Collaboratorive Study Group. AIDS Res Hum Retroviruses. 2000 Aug 10;16(12):1105-11. doi: 10.1089/088922200414947. PMID 10954885
- [Result] Hessol NA, Seaberg EC, Preston-Martin S, Massad LS, Sacks HS, Silver S, Melnick S, Abulafia O, Levine AM; WIHS Collaborative Study Group. Cancer risk among participants in the women's interagency HIV study. J Acquir Immune Defic Syndr. 2004 Aug 1;36(4):978-85. doi: 10.1097/00126334-200408010-00013. PMID 15220706
- [Result] Palacio H, Li X, Wilson TE, Sacks H, Cohen MH, Richardson J, Young M, Munoz A; Women's Interagency HIV Study (WIHS). Healthcare use by varied highly active antiretroviral therapy (HAART) strata: HAART use, discontinuation, and naivety. AIDS. 2004 Mar 5;18(4):621-30. doi: 10.1097/00002030-200403050-00006. PMID 15090767
- [Result] Szczech LA, Hoover DR, Feldman JG, Cohen MH, Gange SJ, Gooze L, Rubin NR, Young MA, Cai X, Shi Q, Gao W, Anastos K. Association between renal disease and outcomes among HIV-infected women receiving or not receiving antiretroviral therapy. Clin Infect Dis. 2004 Oct 15;39(8):1199-206. doi: 10.1086/424013. Epub 2004 Sep 27. PMID 15486845
- [Result] Berhane K, Karim R, Cohen MH, Masri-Lavine L, Young M, Anastos K, Augenbraun M, Watts DH, Levine AM. Impact of highly active antiretroviral therapy on anemia and relationship between anemia and survival in a large cohort of HIV-infected women: Women's Interagency HIV Study. J Acquir Immune Defic Syndr. 2004 Oct 1;37(2):1245-52. doi: 10.1097/01.qai.0000134759.01684.27. PMID 15385731
- [Result] Silverberg MJ, Gore ME, French AL, Gandhi M, Glesby MJ, Kovacs A, Wilson TE, Young MA, Gange SJ. Prevalence of clinical symptoms associated with highly active antiretroviral therapy in the Women's Interagency HIV Study. Clin Infect Dis. 2004 Sep 1;39(5):717-24. doi: 10.1086/423181. Epub 2004 Aug 16. PMID 15356788
- [Result] Tien PC, Cole SR, Williams CM, Li R, Justman JE, Cohen MH, Young M, Rubin N, Augenbraun M, Grunfeld C. Incidence of lipoatrophy and lipohypertrophy in the women's interagency HIV study. J Acquir Immune Defic Syndr. 2003 Dec 15;34(5):461-6. doi: 10.1097/00126334-200312150-00003. PMID 14657755
- [Result] Viscidi RP, Ahdieh-Grant L, Schneider MF, Clayman B, Massad LS, Anastos KM, Burk RD, Minkoff H, Palefsky J, Levine A, Strickler H. Serum immunoglobulin A response to human papillomavirus type 16 virus-like particles in human immunodeficiency virus (HIV)-positive and high-risk HIV-negative women. J Infect Dis. 2003 Dec 15;188(12):1834-44. doi: 10.1086/379975. Epub 2003 Dec 5. PMID 14673762
- [Result] Wilson TE, Barron Y, Cohen M, Richardson J, Greenblatt R, Sacks HS, Young M; Women's Interagency HIV Study. Adherence to antiretroviral therapy and its association with sexual behavior in a national sample of women with human immunodeficiency virus. Clin Infect Dis. 2002 Feb 15;34(4):529-34. doi: 10.1086/338397. Epub 2002 Jan 9. PMID 11797182
- [Result] Wilson TE, Gore ME, Greenblatt R, Cohen M, Minkoff H, Silver S, Robison E, Levine A, Gange SJ. Changes in sexual behavior among HIV-infected women after initiation of HAART. Am J Public Health. 2004 Jul;94(7):1141-6. doi: 10.2105/ajph.94.7.1141. PMID 15226134
- [Result] Ahdieh-Grant L, Li R, Levine AM, Massad LS, Strickler HD, Minkoff H, Moxley M, Palefsky J, Sacks H, Burk RD, Gange SJ. Highly active antiretroviral therapy and cervical squamous intraepithelial lesions in human immunodeficiency virus-positive women. J Natl Cancer Inst. 2004 Jul 21;96(14):1070-6. doi: 10.1093/jnci/djh192. PMID 15265968
- [Result] Anastos K, Barron Y, Cohen MH, Greenblatt RM, Minkoff H, Levine A, Young M, Gange SJ. The prognostic importance of changes in CD4+ cell count and HIV-1 RNA level in women after initiating highly active antiretroviral therapy. Ann Intern Med. 2004 Feb 17;140(4):256-64. doi: 10.7326/0003-4819-140-4-200402170-00007. PMID 14970148
- [Result] Augenbraun M, Goedert JJ, Thomas D, Feldman J, Seaberg EC, French AL, Robison E, Nowicki M, Terrault N. Incident hepatitis C virus in women with human immunodeficiency virus infection. Clin Infect Dis. 2003 Nov 15;37(10):1357-64. doi: 10.1086/379075. Epub 2003 Oct 14. PMID 14583870
- [Result] Barron Y, Cole SR, Greenblatt RM, Cohen MH, Anastos K, DeHovitz JA, Delapenha R, Gange SJ. Effect of discontinuing antiretroviral therapy on survival of women initiated on highly active antiretroviral therapy. AIDS. 2004 Jul 23;18(11):1579-84. doi: 10.1097/01.aids.0000131359.37210.1f. PMID 15238776
- [Result] Cejtin HE, Jacobson L, Springer G, Watts DH, Levine A, Greenblatt R, Anastos K, Minkoff HL, Massad LS, Schmidt JB. Effect of hormonal contraceptive use on plasma HIV-1-RNA levels among HIV-infected women. AIDS. 2003 Jul 25;17(11):1702-4. doi: 10.1097/00002030-200307250-00019. PMID 12853757
- [Result] Cole SR, Hernan MA, Robins JM, Anastos K, Chmiel J, Detels R, Ervin C, Feldman J, Greenblatt R, Kingsley L, Lai S, Young M, Cohen M, Munoz A. Effect of highly active antiretroviral therapy on time to acquired immunodeficiency syndrome or death using marginal structural models. Am J Epidemiol. 2003 Oct 1;158(7):687-94. doi: 10.1093/aje/kwg206. PMID 14507605
- [Result] Falusi O, French AL, Seaberg EC, Tien PC, Watts DH, Minkoff H, Piessens E, Kovacs A, Anastos K, Cohen MH. Prevalence and predictors of Toxoplasma seropositivity in women with and at risk for human immunodeficiency virus infection. Clin Infect Dis. 2002 Dec 1;35(11):1414-7. doi: 10.1086/344462. Epub 2002 Nov 11. PMID 12439806
- [Result] Feldman JG, Gange SJ, Bacchetti P, Cohen M, Young M, Squires KE, Williams C, Goldwasser P, Anastos K. Serum albumin is a powerful predictor of survival among HIV-1-infected women. J Acquir Immune Defic Syndr. 2003 May 1;33(1):66-73. doi: 10.1097/00126334-200305010-00010. PMID 12792357
- [Result] French AL, Benning L, Anastos K, Augenbraun M, Nowicki M, Sathasivam K, Terrault NA. Longitudinal effect of antiretroviral therapy on markers of hepatic toxicity: impact of hepatitis C coinfection. Clin Infect Dis. 2004 Aug 1;39(3):402-10. doi: 10.1086/422142. Epub 2004 Jul 12. PMID 15307009
- [Result] Greenspan D, Gange SJ, Phelan JA, Navazesh M, Alves ME, MacPhail LA, Mulligan R, Greenspan JS. Incidence of oral lesions in HIV-1-infected women: reduction with HAART. J Dent Res. 2004 Feb;83(2):145-50. doi: 10.1177/154405910408300212. PMID 14742653
- [Result] Landay A, Benning L, Bremer J, Weiser B, Burger H, Nowicki M, Kovacs A. Correlates of immune activation marker changes in human immunodeficiency virus (HIV)-seropositive and high-risk HIV-seronegative women who use illicit drugs. J Infect Dis. 2003 Jul 15;188(2):209-18. doi: 10.1086/376509. Epub 2003 Jul 1. PMID 12854075
- [Result] Massad LS, Springer G, Jacobson L, Watts H, Anastos K, Korn A, Cejtin H, Stek A, Young M, Schmidt J, Minkoff H. Pregnancy rates and predictors of conception, miscarriage and abortion in US women with HIV. AIDS. 2004 Jan 23;18(2):281-6. doi: 10.1097/00002030-200401230-00018. PMID 15075546
- [Result] Massad LS, Seaberg EC, Watts DH, Hessol NA, Melnick S, Bitterman P, Anastos K, Silver S, Levine AM, Minkoff H. Low incidence of invasive cervical cancer among HIV-infected US women in a prevention program. AIDS. 2004 Jan 2;18(1):109-13. doi: 10.1097/00002030-200401020-00013. PMID 15090836
- [Result] Navazesh M, Mulligan R, Barron Y, Redford M, Greenspan D, Alves M, Phelan J; Women's Interagency HIV Study participants. A 4-year longitudinal evaluation of xerostomia and salivary gland hypofunction in the Women's Interagency HIV Study participants. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Jun;95(6):693-8. doi: 10.1067/moe.2003.230. PMID 12789150
- [Result] Philpott S, Weiser B, Tarwater P, Vermund SH, Kleeberger CA, Gange SJ, Anastos K, Cohen M, Greenblatt RM, Kovacs A, Minkoff H, Young MA, Miotti P, Dupuis M, Chen CH, Burger H. CC chemokine receptor 5 genotype and susceptibility to transmission of human immunodeficiency virus type 1 in women. J Infect Dis. 2003 Feb 15;187(4):569-75. doi: 10.1086/367995. Epub 2003 Jan 29. PMID 12599073
- [Result] Gandhi M, Ameli N, Bacchetti P, Sharp GB, French AL, Young M, Gange SJ, Anastos K, Holman S, Levine A, Greenblatt RM. Eligibility criteria for HIV clinical trials and generalizability of results: the gap between published reports and study protocols. AIDS. 2005 Nov 4;19(16):1885-96. doi: 10.1097/01.aids.0000189866.67182.f7. PMID 16227797
- [Result] Kovacs A, Wasserman SS, Burns D, Wright DJ, Cohn J, Landay A, Weber K, Cohen M, Levine A, Minkoff H, Miotti P, Palefsky J, Young M, Reichelderfer P; DATRI Study Group; WIHS Study Group. Determinants of HIV-1 shedding in the genital tract of women. Lancet. 2001 Nov 10;358(9293):1593-601. doi: 10.1016/S0140-6736(01)06653-3. PMID 11716886
- [Result] Schneider MF, Gange SJ, Williams CM, Anastos K, Greenblatt RM, Kingsley L, Detels R, Munoz A. Patterns of the hazard of death after AIDS through the evolution of antiretroviral therapy: 1984-2004. AIDS. 2005 Nov 18;19(17):2009-18. doi: 10.1097/01.aids.0000189864.90053.22. PMID 16260908
- [Result] Chu H, Gange SJ, Yamashita TE, Hoover DR, Chmiel JS, Margolick JB, Jacobson LP. Individual variation in CD4 cell count trajectory among human immunodeficiency virus-infected men and women on long-term highly active antiretroviral therapy: an application using a Bayesian random change-point model. Am J Epidemiol. 2005 Oct 15;162(8):787-97. doi: 10.1093/aje/kwi268. Epub 2005 Aug 31. PMID 16135508
- [Result] Ameli N, Bacchetti P, Morrow RA, Hessol NA, Wilkin T, Young M, Cohen M, Minkoff H, Gange SJ, Greenblatt RM. Herpes simplex virus infection in women in the WIHS: epidemiology and effect of antiretroviral therapy on clinical manifestations. AIDS. 2006 Apr 24;20(7):1051-8. doi: 10.1097/01.aids.0000222078.75867.77. PMID 16603858
- [Result] Navazesh M, Mulligan R, Pogoda J, Greenspan D, Alves M, Phelan J, Greenspan J, Slots J. The effect of HAART on salivary microbiota in the Women's Interagency HIV Study (WIHS). Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Dec;100(6):701-8. doi: 10.1016/j.tripleo.2004.10.011. Epub 2005 Jan 25. PMID 16301151
- [Result] Liu C, Weber K, Robison E, Hu Z, Jacobson LP, Gange SJ. Assessing the effect of HAART on change in quality of life among HIV-infected women. AIDS Res Ther. 2006 Mar 20;3:6. doi: 10.1186/1742-6405-3-6. PMID 16549012
- [Derived] Haley DF, Bullington BW, Tien P, Knittel AK, Bobitt J, Kempf MC, Philbin M, Hanna DB, Lindsey S, Kassaye S, DeHovitz J, Cohen M, Wingood G, Jones DL, Williams MP, Wang RJ, Edmonds A. Patterns of Cannabis Use among Women With HIV in the United States. AIDS Behav. 2025 Jun;29(6):2022-2032. doi: 10.1007/s10461-025-04669-z. Epub 2025 Mar 7. PMID 40050488
- [Derived] Daubert EM, Dionne J, Atrio J, Knittel AK, Kassaye SG, Seidman D, Long A, Brockmann S, Ofotokun I, Fischl MA, Massad LS, Weber KM. Declining Prevalence of Trichomonas vaginalis Diagnosed by Wet Mount in a Cohort of U.S. Women With and Without HIV. J Womens Health (Larchmt). 2024 Mar;33(3):388-395. doi: 10.1089/jwh.2023.0263. Epub 2024 Jan 12. PMID 38215275
- [Derived] Cohen MH, Benning L, Weber KM, Sharma A, Plankey M, Kempf MC, Wilson TE, Aouizerat B, Milam J, Adimora AA, Wingood G, Carrico AW. Predictors and Consequences of Prescription Opioid Use in Women Living With and Without HIV: 20-Year Follow-Up. J Womens Health (Larchmt). 2022 Aug;31(8):1188-1196. doi: 10.1089/jwh.2021.0231. Epub 2022 Feb 28. PMID 35230165
- [Derived] Massad LS, Daubert EM, Evans CT, Minkoff H, Kassaye S, Dionne-Odom J, Seidman D, Murphy K, Alcaide ML, Adimora AA, Sheth AN, Golub ET, French AL, Weber KM. Trends in Bacterial Vaginosis Prevalence in a Cohort of U.S. Women with and at Risk for HIV. J Womens Health (Larchmt). 2022 May;31(5):726-732. doi: 10.1089/jwh.2021.0102. Epub 2021 Aug 27. PMID 34449258
- [Derived] Kato Y, Kizer JR, Ostovaneh MR, Lazar J, Peng Q, van der Geest RJ, Lima JAC, Ambale-Venkatesh B. Extracellular volume-guided late gadolinium enhancement analysis for non-ischemic cardiomyopathy: The Women's Interagency HIV Study. BMC Med Imaging. 2021 Jul 27;21(1):116. doi: 10.1186/s12880-021-00649-6. PMID 34315432
- [Derived] Haley DF, Edmonds A, Ramirez C, French AL, Tien P, Thio CL, Witt MD, Seaberg EC, Plankey MW, Cohen MH, Adimora AA. Direct-Acting Antiviral Hepatitis C Treatment Cascade and Barriers to Treatment Initiation Among US Men and Women With and Without HIV. J Infect Dis. 2021 Jun 15;223(12):2136-2144. doi: 10.1093/infdis/jiaa686. PMID 33141170
- [Derived] Haley DF, Kramer MR, Adimora AA, Haardorfer R, Wingood GM, Ludema C, Rubtsova A, Hickson DA, Ross Z, Golub E, Bolivar H, Cooper HL. Relationships between neighbourhood characteristics and current STI status among HIV-infected and HIV-uninfected women living in the Southern USA: a cross-sectional multilevel analysis. Sex Transm Infect. 2017 Dec;93(8):583-589. doi: 10.1136/sextrans-2016-052889. Epub 2017 Mar 7. PMID 28270536
- [Derived] Massad LS, Xie X, Darragh T, Minkoff H, Levine AM, Watts DH, Wright RL, D'Souza G, Colie C, Strickler HD; Women's Interagency HIV Study Collaborative Study Group. Genital warts and vulvar intraepithelial neoplasia: natural history and effects of treatment and human immunodeficiency virus infection. Obstet Gynecol. 2011 Oct;118(4):831-9. doi: 10.1097/AOG.0b013e31821a0f4d. PMID 21934446
- See also: Click here for the WIHS homepage. — http://statepiaps.jhsph.edu/wihs/